CLINICAL TRIAL: NCT02115893
Title: The Effect of Nitrate Supplementation on Sports Performance: Duration of Supplementation
Brief Title: Nitrate Supplementation; Duration
Acronym: NO-how
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: METC13-3-059
Record Dates: First submitted 2014-04-10; First posted 2014-04-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2014-10

CONDITIONS: Time-trial Performance; Submaximal Exercise Performance; Nitrite; Nitrate
Keywords: Nitrate; Performance; Sports
MeSH Terms: interventions — sodium nitrate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sodium Nitrate (Active Comparator): Dietary Supplement: Sodium nitrate 800 mg of nitrate in sodium nitrate added with water to get a 140 mL solution (BASF, Ludwigshafen, Germany)
  Interventions: Dietary Supplement: Sodium Nitrate
- Sodium Cloride (Placebo Comparator): Dietary Supplement: Sodium chloride 800 mg of sodium chloride added with water to get a 140 mL solution (Frisia Zout BV, Harlingen, The Netherlands)
  Interventions: Dietary Supplement: Sodium Chloride

INTERVENTIONS:
Dietary Supplement: Sodium Nitrate
  Arms: Sodium Nitrate
Dietary Supplement: Sodium Chloride
  Arms: Sodium Cloride

SUMMARY:
The main aim of the current study will be to find the optimal duration of supplementation to enhance sports performance.

DETAILED DESCRIPTION:
Oral ingestion of nitrate (NO3-) in the form of both nitrate salts and beetroot juice has been shown to significantly lower blood pressure at rest and to also lower pulmonary oxygen uptake during exercise, in addition to improving exercise performance during cycle time trial. However, there has been no consensus on the optimal supplementation protocols, in terms of duration of supplementation to see these metabolic effects. Furthermore, a positive exercise performance effect of nitrate ingestion has primarily been observed in recreational athletes. The potentially ergogenic effects of nitrate in well-trained or elite athletes therefore remain to be fully established. Based on the gaps in current literature, our main goal will be to gain further insight into different aspects of nitrate supplementation to enhance (elite) sports performance. This will be investigated in this study by assessing the effect of an acute vs. chronic supplementation period of sodium nitrate (NaNO3-) on exercise performance.

ELIGIBILITY:
Inclusion Criteria:

* 18.5 < BMI < 25 kg/m2
* Endurance trained cyclists/triathletes (with at least 1 year of competitive cycling experience)
* VO2max ≥ 55 mL/kg/min

Exclusion Criteria:

* Use of medication
* Injury prohibiting them from performing the exercise protocol effectively
* Smoking
* Currently supplementing diet with nitrate
* Lactose intolerance

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2014-11 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Time-trial exercise performance | Time trial starts 4 hours after ingestion and ends on average after 15 minutes of cycling (depending on subject's cycling speed)
  The primary outcome measure will be the time to complete the time-trial following dietary nitrate or placebo ingestion

SECONDARY OUTCOMES:
Resting blood pressure | 30 min pre-ingestion until 2.5 hours post-ingestion
  Resting blood pressure measures following ingestion of dietary nitrate
Plasma nitrate and nitrite levels | 30 min pre-ingestion until 30 min post-time-trial testing
  Plasma nitrate and nitrite levels following ingestion of dietary nitrate
Submaximal exercise performance | starting from 3 hours post-ingestion on testing days until completion of the submaximal exercise
  Oxygen consumption CO2 production and heart rate during submaximal exercise
Time-trial exercise performance; power output and heart rate | starting from 4 hours post-ingestion on testing days until completion of the time-trial
  Power output and heart rate during the time-trial exercise

OTHER OUTCOMES:
Baseline characteristics and fitness level assessment | 3 hours during visit 1 (Screening)
  Resting blood pressure, height, body weight, age, BMI, measures of GI tolerance, VO2 max, Wmax, rate of perceived exertion

CONTACTS AND LOCATIONS:
Overall Officials: Lex B Verdijk, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Centre+, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Wylie LJ, Kelly J, Bailey SJ, Blackwell JR, Skiba PF, Winyard PG, Jeukendrup AE, Vanhatalo A, Jones AM. Beetroot juice and exercise: pharmacodynamic and dose-response relationships. J Appl Physiol (1985). 2013 Aug 1;115(3):325-36. doi: 10.1152/japplphysiol.00372.2013. Epub 2013 May 2. PMID 23640589
- [Background] Cermak NM, Gibala MJ, van Loon LJ. Nitrate supplementation's improvement of 10-km time-trial performance in trained cyclists. Int J Sport Nutr Exerc Metab. 2012 Feb;22(1):64-71. doi: 10.1123/ijsnem.22.1.64. PMID 22248502
- [Background] Bescos R, Sureda A, Tur JA, Pons A. The effect of nitric-oxide-related supplements on human performance. Sports Med. 2012 Feb 1;42(2):99-117. doi: 10.2165/11596860-000000000-00000. PMID 22260513